CLINICAL TRIAL: NCT01617746
Title: Examination of the Bronchoprotective Effect of Endothelin Receptor Blockade in Asthma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Mark Spears, Clinical Lecturer, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR012
Record Dates: First submitted 2012-03-07; First posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Asthma
Keywords: Asthma; Endothelin; Airway hyperreactivity
MeSH Terms: conditions — Asthma | interventions — ambrisentan; Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ambrisentan (Experimental): 5mg od ambrisentan
  Interventions: Drug: Ambrisentan
- Bosentan (Experimental): 62.5mg bosentan
  Interventions: Drug: Bosentan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ambrisentan — 5mg od two weeks
  Other Names: Volibris
  Arms: Ambrisentan
Drug: Bosentan — 62.5mg bd two weeks
  Other Names: Tracleer
  Arms: Bosentan
Drug: Placebo — bd for two weeks
  Arms: Placebo

SUMMARY:
The purpose of this study will be to determine if blockade of endothelin 1 signalling via endothelin receptor A using ambrisentan or dual blockade (A&B) via bosentan can provide protection against methacholine induced bronchoconstriction in asthma.

DETAILED DESCRIPTION:
Endothelin 1 may have a role in the development of acute airway narrowing in asthma. Blockade of the endothelin system may thereby protect against airway narrowing. Two receptors exist for endothelin 1, Endothelin A & B. Both can be blocked by Bosentan, and the A receptor by ambrisentan. Both medications are currently in use for the treatment of pulmonary arterial hypertension. The investigators will endeavour to examine the potential role of endothelin 1 in the development of airway narrowing in asthma through blockade of the endothelin receptors A&B through the use of bosentan and ambrisentan.

ELIGIBILITY:
Inclusion Criteria:

1. Physician diagnosis of asthma confirmed objectively by airway hyperactivity to methacholine (as determined by a ≥ 20% drop in FEV at a methacholine dose of ≤ 8mg/ml after β-agonist withdrawal as per ATS guidelines)
2. Age range 18-60 years
3. FEV1 ≥ 60% predicted
4. Duration of asthma > 6 months and on stable medication for 4 weeks
5. Prescribed and compliant with inhaled corticosteroid up to a maximum of 2000mcg beclomethasone or equivalent
6. No history of previous regular smoking and current non-smoker

Exclusion Criteria:

1. Unstable asthma; defined as the presence of 1 or more of the following events in the month prior to study [Emergency/'out of hours' visit to GP for asthma exacerbation; GP visit to patient at home for asthma exacerbation or A & E/hospital admission for asthma exacerbation]
2. Treatment with oral corticosteroids in the past month
3. Need for maintenance oral corticosteroid therapy
4. Pregnancy or planning to become pregnant over course of study and up to one month after
5. Excessive risk of hepatotoxicity from endothelin receptor antagonists;

   * Alcohol excess (defined as regular consumption above government daily recommend limits; currently defined as 28 units per wk for men, 21 units per week for women)
   * Previous intravenous drug use
   * Current or known history of liver disease (with the exception of Gilberts disease and gallstones)
   * Chronic hepatitis (either viral (e.g. hepatitis B or C) or autoimmune)
   * Bilirubin, alanine aminotransferase (ALT) or asparate aminotransferase (AST) greater than the upper limit of normal at screening
6. Anaemia (defined as haemoglobin below the lower reference range for sex) at screening
7. Renal failure (defined as eGFR less than 50 mL/minute/1.73 m2) at screening
8. Known HIV positivity
9. History of inability to tolerate bosentan or ambrisentan
10. Significant medical conditions other than asthma felt by investigator to preclude participation in study. This could be either in patients best interest or due to potential to significantly alter responses to medication and hence alter power of clinical trial (examples include; significant heart failure (NYHA grades II-IV), diabetes mellitus, bronchiectasis or haematological malignancy).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Difference in doubling dose of methacholine to produce bronchoconstriction compared to placebo | 2 weeks
  Both active treatments will be compared against placebo with respect to protection against methacholine induced bronchoconstriction

SECONDARY OUTCOMES:
Which of the endothelin receptors A&B are most bronchoprotective against methacholine | 2 weeks
  Both bostentan and ambrisentans effect on airway response to methacholine will be compared to placebo. The relative efficacy will be compared, in terms of doubling doses of methacholine.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Spears, MBChB PhD, Principal Investigator — University of Glasgow
Locations (1):
- Asthma Research Unit, University of Glasgow, Glasgow, United Kingdom